CLINICAL TRIAL: NCT04601857
Title: A Phase 2 Study Evaluating Futibatinib (TAS 120) Plus Pembrolizumab in the Treatment of Advanced or Metastatic Urothelial Carcinoma
Brief Title: Futibatinib and Pembrolizumab Combination in the Treatment of Advanced or Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to discontinue the study due to strategic considerations and not due to any safety-related concerns.
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-203; 2020-000945-15 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-26 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Advanced and Metastatic Urothelial Cancer
Keywords: Futibatinib; Pembrolizumab; Urothelial cancer; FGFR; TAS120; MK3475 B04
MeSH Terms: interventions — futibatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants with metastatic urothelial carcinoma (UC) and FGFR3 mutation or FGFR1-4 fusion/rearrangement received futibatinib 20 milligrams (mg), orally, once daily (QD), in a 21-day cycle for maximum duration of 590 days along with pembrolizumab 200 mg, intravenously (IV), every 3 weeks (Q3W), in a 21-day cycle for a maximum of 35 doses or a maximum duration of 2 years.
  Interventions: Drug: Futibatinib; Drug: Pembrolizumab
- Cohort B (Experimental): Participants with metastatic UC (including participants with other FGFR or non-FGFR genetic aberrations and participants with wild type [non-mutated] tumors) received futibatinib 20 mg, orally, QD, in a 21-day cycle for maximum duration of 563 days along with pembrolizumab 200 mg, IV, Q3W in a 21-day cycle for a maximum of 35 doses or a maximum duration of 2 years.
  Interventions: Drug: Futibatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Futibatinib — Oral
  Other Names: TAS120
Drug: Pembrolizumab — IV
  Other Names: KEYTRUDA; MK-3475-B04

SUMMARY:
The purpose of the trial is to evaluate the antitumor activity and confirm the safety for the combination of Fibroblast Growth Factor Receptor (FGFR) inhibitor futibatinib and anti-programmed cell death-1 (PD-1) antibody pembrolizumab in patients with advanced or metastatic urothelial cancer who are not candidates to receive a platinum-based treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. Age ≥ 18 years of age
3. Histologically confirmed advanced or metastatic urothelial carcinoma who have not received systemic treatment for advanced metastatic disease.

   1. Cohort A: must have an FGFR3 mutation or FGFR1-4 fusion/rearrangement.
   2. Cohort B: all other patients with UC (including patients with other FGFR or non-FGFR genetic aberrations and patients with wild-type [non-mutated] tumors)
4. Unfit for or intolerant to standard platinum-based chemotherapy.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1.
6. Adequate organ function.
7. Have a measurable disease per RECIST 1.1

Exclusion Criteria:

1. Have received prior therapy with anti-PD-1, anti-PD-L1/L2 agent or FGFR inhibitor.
2. History and/or current evidence of any of the following disorders:

   1. Non-tumor related alteration of the calcium-phosphorus homeostasis that is considered clinically significant in the opinion of the Investigator.
   2. Ectopic mineralization/calcification considered clinically significant in the opinion of the Investigator.
   3. Retinal or corneal disorder considered clinically significant in the opinion of the Investigator.
3. Has received a live vaccine within 30 days prior to the first dose of study drug.
4. Have an active autoimmune disease that has required systemic treatment in the past 2 years.
5. Have a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
6. Have had an allogenic tissue/ organ transplant.
7. Has known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA.
8. Have known active central nervous system metastases and/or carcinomatous meningitis.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2025-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Care Centers of Nevada, Las Vegas, Nevada
- France (6):
  - ICANS - Institut de cancérologie de Strasbourg Europe, Strasbourg, Bas-Rhin
  - Institut Paoli Calmettes - HÃ´pital de jour, Marseille, Bouches-du-Rhône
  - Centre Georges-François Leclerc, Dijon, Côte d'Or
  - Centre Leon Berard - departement d'oncologie medicale, Lyon, Rhone
  - Centre Regional de Lutte Contre le Cancer de Lorraine, Vandœuvre-lès-Nancy
  - Institut De Cancerologie Gustave Roussy, Villejuif
- Spain (8):
  - ALTHAIA, Xarxa Assistencial Universitària de Manresa, Manresa, Brcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario HMN Sanchinarro, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 sites in the United States, France and Spain from 07 January 2021 to 16 September 2025.
Pre-assignment Details: A total of 43 participants were enrolled to receive futibatinib along with pembrolizumab.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 17 | 26
Completed | 5 | 1
Not Completed | 12 | 25
Not completed — Adverse Event/Serious Adverse Event | 3 | 7
Not completed — Disease Progression | 2 | 4
Not completed — Clinical Disease Progression | 2 | 1
Not completed — Radiological Progression | 4 | 11
Not completed — Death | 1 | 0
Not completed — Reason Not Specified | 0 | 1
Not completed — At the Participant's Request | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated population included all participants in all enrolled population who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 17 | 26 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (9.86) | 72.2 (10.03) | 72.6 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 14 | 23 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 7 | 17 | 24
  Unknown or Not Reported | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 1 | 1 | 2
  Caucasian/White | 7 | 15 | 22
  Other | 0 | 1 | 1
  Not Reported | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants experiencing a best overall response of partial response (PR) or complete response (CR) according to response evaluation criteria in solid tumors, version 1.1 (RECIST 1.1) criteria based on investigator assessment. Evaluation of target lesions defined a CR as the disappearance of all target lesions and non-target lesions (if applicable), and normalization of tumor marker level; PR was defined as at least a 30 percent (%) decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum of diameters for all target lesion assessments. Evaluation of non-target lesions was defined as the persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. For both target and non-target evaluations, any pathological lymph node must have had a reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: Up to 38 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 26
percentage of participants | 47.1 [23.0 to 72.2] | 26.9 [11.6 to 47.8]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants experiencing a best overall response of SD, PR, or CR. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), referencing the smallest sum diameters while on study. Evaluation of target lesions defined a CR as the disappearance of all target lesions and non-target lesions (if applicable), and normalization of tumor marker level; PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum of diameters for all target lesion assessments. Evaluation of non-target lesions was defined as the persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. For both target and non-target evaluations, any pathological lymph node must have had a reduction in short axis <10 mm.
Time Frame: Up to 38 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 26
percentage of participants | 82.4 [56.6 to 96.2] | 53.8 [33.4 to 73.4]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was calculated for all responders from the date of first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause, whichever occurred first. Evaluation of target lesions defined a CR as the disappearance of all target lesions and non-target lesions (if applicable), and normalization of tumor marker level; PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum of diameters for all target lesion assessments. Evaluation of non-target lesions was defined as the persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. For both target and non-target evaluations, any pathological lymph node must have had a reduction in short axis to <10 mm.
Time Frame: Up to 38 months
Population: All treated population included all participants in all enrolled population who received at least one dose of study drug. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 8 | 7
months | 12.32 [6.5 to 24.0] | 14.46 [3.0 to 23.5]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose of study therapy to the date of death (any cause) or disease progression, whichever occurred first. The PFS was analyzed using a Kaplan-Meier method, with PFS time being censored on the date of the last tumor assessment. The 95% confidence interval (CI) for median PFS was provided using the Kaplan-Meier procedure.
Time Frame: Up to 38 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 26
months | 8.3 [3.5 to 18.5] | 4.1 [2.1 to 8.3]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose to the death date. Participants without a documented death date were censored on the last date they were known to be alive.
Time Frame: Up to 38 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 26
months | 16.2 [6.6 to NA] — The upper limit of the 95% CI could not be estimated, as participants were still alive at the data cut-off. | 18.3 [6.2 to NA] — The upper limit of the 95% CI could not be estimated, as participants were still alive at the data cut-off.

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant and does not necessarily have a causal relationship with the study drug. TEAEs are defined as AEs reported up to 30 days after the last dose of any study therapy (safety follow-up) or until the start of new antitumor therapy, whichever is earlier, unless otherwise specified.
Time Frame: Up to 38 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 26
Participants | 17 | 26

ADVERSE EVENTS:
Time Frame: Up to 38 months
Description: All treated population included all participants in all enrolled population who received at least one dose of study drug.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 7/17 | 13/26
Serious Adverse Events (participants affected / at risk) | 10/17 | 12/26
Other Adverse Events (participants affected / at risk) | 17/17 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=17) | Cohort B (N=26)
Cardiac tamponade (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
General physical health deterioration (General disorders) | 2 | 3
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Urethral fistula (Renal and urinary disorders) | 0 | 1
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=17) | Cohort B (N=26)
Anaemia (Blood and lymphatic system disorders) | 7 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Conduction disorder (Cardiac disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1
Immune-mediated hyperthyroidism (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 3 | 2
Vision blurred (Eye disorders) | 2 | 2
Central serous chorioretinopathy (Eye disorders) | 1 | 1
Keratitis (Eye disorders) | 1 | 0
Keratopathy (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 1
Macular detachment (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 1 | 0
Vitreous adhesions (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 14
Dry mouth (Gastrointestinal disorders) | 9 | 8
Nausea (Gastrointestinal disorders) | 3 | 9
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Stomatitis (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 8 | 9
Oedema peripheral (General disorders) | 5 | 4
Fatigue (General disorders) | 4 | 7
Mucosal inflammation (General disorders) | 3 | 8
Xerosis (General disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 3 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Paronychia (Infections and infestations) | 3 | 1
Oral fungal infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 2
Otitis externa fungal (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 4
COVID-19 (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 7 | 3
Weight decreased (Investigations) | 5 | 9
Blood alkaline phosphatase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 5
Alanine aminotransferase increased (Investigations) | 2 | 4
Blood triglycerides increased (Investigations) | 2 | 0
Blood albumin increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Capillary nail refill test abnormal (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 12 | 13
Decreased appetite (Metabolism and nutrition disorders) | 9 | 13
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Cell death (Metabolism and nutrition disorders) | 1 | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Dysgeusia (Nervous system disorders) | 5 | 8
Aphasia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Testicular oedema (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 3 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 1
Anhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 1 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Yellow nail syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04601857/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04601857/SAP_001.pdf